CLINICAL TRIAL: NCT04920734
Title: Description of Therapy Options and Successes in the Long-term Course of Delirium in the Recovery Room - Multicenter Observational Study (CESARO-2)
Brief Title: Description of Therapy Options and Successes in the Long-term Course of Delirium in the Recovery Room - CESARO II
Status: Terminated | Type: Observational
Why Stopped: Lack of equipment
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ.- Prof. Dr. C. Spies, Charite University, Berlin, Germany
Other Study IDs: CESARO-2
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a multicenter pilot project to evaluate the therapeutic success in the long term up to 3 months after a delirium in a recovery room. There is a Europe-wide recommendation for the prevention of postoperative delirium in older patients and the evidence and consensus-based guideline "Management of delirium, analgesia and sedation in intensiv care medicine" of the AWMF (Arbeitsgemeinschaft der Wissenschaftlichen Medizinischen Fachgesellschaften) are regularly updated for the detection and treatment of delirium in the intensive care unit. The aim is to evaluate the effects of a systematic delirium screening and the delirium treatment options in the long term in the same way as the current recommendations for the patient cohort of the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the recovery room who have been diagnosed with delirium according to the treating physicians
* The patient is on a ward in the hospital
* Age ≥ 18 years
* Stay in the recovery room ≥ 1 day
* The patient is able to give consent

Exclusion Criteria:

* Participation in a prospective intervention study (except adjuvant therapy study)
* Patients with underlying neurological diseases that make it difficult to differentiate from delirium
* Missing contact 3 months after stay in the recovery room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the recovery room who have been diagnosed with delirium
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Morbidity | Up to three months
  Postoperative complications according to Clavien-Dindo classification

SECONDARY OUTCOMES:
Duration of delirium | Time until discharge from recovery room, an expected average of 5 days
  Duration of delirium is measured in days
Incidence of delirium | Time until discharge from recovery room, an expected average of 5 days
  Postoperative delirium rate, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) and/or as ≥ 2 cumulative points in the Nursing Delirium Screening Scale (Nu-DESC) and/or a positive Confusion Assessment Method (CAM) and/or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score and/or patient chart review that shows descriptions of delirium.
Preventive measures against delirium 1 | Time until discharge from recovery room, an expected average of 5 days
  Preventive measures of delirium are measured by medical treatments
Preventive measures against delirium 2 | Time until discharge from recovery room, an expected average of 5 days
  Preventive measures of delirium are measured by non-medical treatments
Anticholinergic drugs | Time until discharge from hospital, an expected average of 7 days
  Measured by anticholinergic drug scale
Treatment of delirium | Time until discharge from hospital, an expected average of 7 days
  Treatment of delirium with medication
Measurement of acetylcholinesterase | Time until discharge from recovery room, an expected average of 5 days
  Measurement of activities of the enzyme - acetylcholinesterase in blood
Measurement of butyrylcholinesterase | Time until discharge from recovery room, an expected average of 5 days
  Measurement of activities of the enzyme - butyrylcholinesterase in blood
Chronic comorbid diseases | Time until discharge from hospital, an expected average of 7 days
  Chronic comorbid diseases (comorbidities) are measured by Charlson comorbidity index
Health related quality of life | Up to three months
  EQ-5D
Treatment of vegetative symptoms | Time until discharge from recovery room, an expected average of 5 days
  Treatment of vegetative symptoms is measured by vegetative medical therapy
Treatment of pain | Time until discharge from recovery room, an expected average of 5 days
  Treatment of pain is measured by analgesia
Treatment of postoperative vomiting | Time until discharge from recovery room, an expected average of 5 days
  Treatment of postoperative vomiting is measured by anti-emetics
Treatment of productive psychotic symptoms | Time until discharge from recovery room, an expected average of 5 days
  Treatment of productive psychotic symptoms is measured by anti-psychotics
Treatment of anxiety | Time until discharge from recovery room, an expected average of 5 days
  Treatment of anxiety is measured by anxiolytics
Treatment of sleep disorders | Time until discharge from recovery room, an expected average of 5 days
  Treatment of sleep disorders are measured by sleeping drugs
Number of participants with changes in laboratory values | Time until discharge from hospital, an expected average of 7 days
  Routine laboratory results were planned to be documented in the hospital including hemoglobin, lymphocytes, total neutrophils, platelet count and white blood cell (WBC) count from blood samples.
Apache II | Time until discharge from intensive care unit, an expected average of 6 days
  APACHE II score is measured by the Acute Physiology and Chronic Health Evaluation System II.
SOFA | Time until discharge from intensive care unit, an expected average of 6 days
  SOFA is measured by Sequential Organ Failure Assessment.
SAPS II | Time until discharge from intensive care unit, an expected average of 6 days
  SAPS II is measured by Simplified Acute Physiology Score II.
Intensive care unit stay | Time until discharge from intensive care unit, an expected average of 6 days
  Intensive care unit stay is measured in days
Hospital stay | Time until discharge from hospital, an expected average of 7 days
  Hospital stay is measured in days

OTHER OUTCOMES:
Patient-specific characteristics | At the beginning of the investigation
  Patient-specific characteristics are measured by demographic data

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No